CLINICAL TRIAL: NCT02593864
Title: A Novel Serum Biomarker Stress Test for Detection of Early Osteoarthritis
Brief Title: A Biomarker Stress Test for Detection of Early Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Constance Chu, MD, Director, Joint Preservation Center, VA Palo Alto Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1I21RX002045 (NIH)
Record Dates: First submitted 2015-10-28; First posted 2015-11-02 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Variable-Stiffness Shoe (Experimental): Subjects will wear a load-modifying variable-stiffness shoe for 6 months
  Interventions: Device: Variable-Stiffness Shoe

INTERVENTIONS:
Device: Variable-Stiffness Shoe — A load-modifying variable-stiffness shoe previously shown to reduce joint loading

SUMMARY:
Veterans have much higher risk of osteoarthritis (OA) then the general population. Knee OA is common among Veterans and is a leading cause of disability. The earliest stages of OA development, where the joint cartilage wears away, is usually painless. By the time Veterans experience symptoms, the OA is typically advanced and there is nothing that can be done except palliation until the joint is replaced with metal and plastic. If there was a blood test to provide early warning of cartilage wear and joint deterioration, Veterans could potentially be treated early enough to slow down or even prevent OA. So far, development of such a blood test has proved elusive. The investigators propose a new method to amplify the signs of cartilage wear in the blood by challenging the affected joint with a walking task. Similar to a cardiac stress test, this walking challenge may help to separate joints at risk from healthy joints. The investigators will also see if this 'OA stress test' can show if a simple and inexpensive load-modifying shoe can improve joint health in Veterans with early knee OA.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* symptomatic medial compartment knee OA (KL grades 0-2)
* full weight-bearing status
* able to walk for 30 minutes or longer
* able to undergo MRI scan
* agreement and ability to use provided shoe as primary walking shoe (4 or more hours a day) during the 6 month study period

Exclusion Criteria:

* inflammatory arthritis, gout or recurrent pseudogout
* patellofemoral or lateral compartment disease that is equal to or more extensive than medial disease
* symptomatic OA of other lower extremity joints
* BMI >35 kg/m2
* prior structural surgery of the knee except for medial meniscectomy performed > 6 months prior
* use of shoe insert or hinged knee brace
* pes planus, and/or unusual foot size or shape

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance Chu, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: X-ray screening for inclusion/exclusion criteria
Period: Overall Study
Arm/Group | Variable-Stiffness Shoe
Started | 25
Completed | 19
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Participants assigned to the variable-stiffness shoe
Arm/Group | Variable-Stiffness Shoe
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Knee Adduction Moment [Mean (Standard Deviation); unit: %Bw*Ht] — Knee adduction moment describes the medial/lateral load distribution of the knee measured while walking in a gait laboratory. Before normalization to account for size, the knee adduction moment is expressed in Nm. However, to account for different sized people, the knee adduction moment is transformed and expressed in percentage of body weight times height (%BW*ht). Population: Per protocol cohort. Baseline value of subjects who completed the 6 month study visit. Gait data unusable for 1 subject at follow-up, and this subject was not included in the baseline value.
  %Bw*Ht
    number analyzed (Participants) | 18
    (all) | 2.67 (0.76)
COMP at 3.5 Hours (% Of Baseline Resting) [Mean (Standard Deviation); unit: % Of Resting] — Serum samples were collected before and after a 30 minute walking activity. Levels of serum cartilage oligomeric matrix protein (COMP) 3.5 hours following the 30-minute walk, expressed as a percentage of pre-activity resting values, were assessed. Population: Per protocol cohort. These analyses are based on available data from 15 subjects who completed both the baseline and follow-up visits for analysis of changes in COMP. Biomarker data for one subject was missing at baseline, and complete biomarker data for 3 subjects was unable to be collected at follow-up.
  % Of Resting
    number analyzed (Participants) | 15
    (all) | 84.4 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: Change at 6 Months From Baseline in First Peak Knee Adduction Moment (KAM): (6 Month Value - Baseline)
Description: Knee adduction moment describes the medial/lateral load distribution of the knee measured while walking in a gait laboratory. Before normalization to account for size, the knee adduction moment is expressed in Nm. However, to account for different sized people, the knee adduction moment is transformed and expressed in percentage of body weight times height (%BW*ht). Higher knee adduction moments have been linked to more severe osteoarthritis (OA). Knee adduction moment will be analyzed at baseline and after 6 months of variable-stiffness shoe wear. Values at 6 months (in variable-stiffness shoe) will be compared to baseline (in control shoe).
Time Frame: Baseline to 6 months
Population: These results were based on gait data for 18 subjects that was available at both the baseline and follow-up visits
Measure: Mean (Standard Deviation); unit: %Bw*Ht
Arm/Group | Variable-Stiffness Shoe
Number analyzed (Participants) | 18
%Bw*Ht | -0.19 (0.17)

2. Primary Outcome: Change at 6 Months From Baseline in Serum COMP Biomarker Levels in Response to a Mechanical Stimulus (6 Month - Baseline)
Description: Serum samples were collected before and after a 30 minute walking activity. Levels of serum cartilage oligomeric matrix protein (COMP) 3.5 hours following the 30-minute walk, expressed as a percentage of pre-activity resting values, were assessed, and values at 6 months were compared to baseline.
Time Frame: Baseline to 6 months
Population: These analyses were based on available data from 15 subjects at both the baseline and follow-up visits for analysis of changes in COMP
Measure: Mean (Standard Deviation); unit: Percent of Resting
Arm/Group | Variable-Stiffness Shoe
Number analyzed (Participants) | 15
Percent of Resting | -0.8 (10.3)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Variable-Stiffness Shoe
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 7/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Variable-Stiffness Shoe (N=25)
Joint paint (Musculoskeletal and connective tissue disorders) | 7 (8) — Related and Un-related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02593864/Prot_SAP_000.pdf